CLINICAL TRIAL: NCT07161375
Title: Infrared Thermography for Prediction of Successful Erector Spinae Plane Block in Unilateral Inguinal Hernia Surgery in Paediatric Patients: A Prospective Observational Study
Brief Title: Infrared Thermography for Prediction of Successful Erector Spinae Plane Block in Unilateral Inguinal Hernia Surgery in Paediatric Patients
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Abdelfatah Abdelrahman Abdelfatah, Assistant Lecturer of Anesthesia, Pain Management and surgical ICU, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Other Study IDs: MD-210-2024
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Infrared; Thermography; Prediction; Erector Spinae Plane Block; Unilateral Inguinal Hernia Surgery; Paediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Children undergoing elective unilateral open inguinal hernia surgery.
  Interventions: Device: Infrared Thermography

INTERVENTIONS:
Device: Infrared Thermography — Infrared thermography will be used to predict the success of an erector spinae block by measuring the temperature difference between the blocked and unblocked sides.

SUMMARY:
This study aims to evaluate the accuracy of temperature change (ΔT) measurements using infrared thermography to predict a successful erector spinae plane block in pediatric patients undergoing inguinal hernia repair under general anesthesia.

DETAILED DESCRIPTION:
Lower abdominal surgeries, including inguinal hernia repair, have been performed extensively in the daily practice of pediatric surgeries, so ensuring sufficient intra- and post-operative analgesia is crucial for perioperative care.

The ultrasound-guided erector spinae plane block (ESPB) is a regional anesthetic technique. Early detection of successful ESPB in pediatric patients will enable the application of rescue techniques at the appropriate time, thereby improving patient satisfaction and reducing operating theatre time.

There is considerable evidence regarding the value of infrared thermography in predicting successful nerve blocks. Infrared thermography is the process of using a thermal image to detect radiation (heat) coming from an object, converting it to temperature, and displaying an image of the temperature distribution.

ELIGIBILITY:
Inclusion Criteria:

* Age from 3 months to 6 years.
* Both genders.
* American Society of Anesthesiologists (ASA) Physical Status I-II.
* Children undergoing elective unilateral open inguinal hernia surgery.

Exclusion Criteria:

* Parents' or guardians' refusal
* Known Allergy to local anesthetics.
* Coagulopathy [international normalised ratio (INR) >1.4 or platelets <75.000].
* Infection at the site of injection or wound close to the puncture site.
* preexisting neuropathy (with sensory and/or motor deficits).
* Diseases interfere with thermal imaging (as skin infections).
* Baseline oesophageal body temperature of more than 37.5 °C.
* Emergency and re-do cases will be excluded.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted at Kasr Al Ainy, Abu El Reesh children hospital.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Predict successful ESPB | Throughout 20 minutes of block
  The ability to predict a successful erector spinae plane block by infrared thermography through the change in temperature (ΔT) (degrees Celsius) between the blocked and unblocked sides of the same dermatomal level in the mid-clavicular line throughout 20 minutes of block.

SECONDARY OUTCOMES:
Degree of pain | 12 hours after surgery
  Degree of pain will be assessed using Face, Legs, Activity, Cry, and Consolability (FLACC) score. Each category is scored from 0 to 2, resulting in a total pain score from 0 to 10, where 0 indicates no pain and higher scores represent increasing pain levels. FLACC will be recorded at 15, 30, 45 and 60 min, 6 and 12 hours after surgery.
Heart rate | Till discharge of the patient (Up to 12 hours)
  Heart rate will be recorded 5 min after intubation, then every 5 min after block 5,10,15, and 20 min, then at skin incision, immediately after extubation, 15 min after extubation, and every 15 minutes in the post-anesthesia care unit (PACU) (30,45, and 60 minutes) till discharge of the patient.
Systolic blood pressure | Till discharge of the patient (Up to 12 hours)
  Systolic blood pressure will be recorded 5 min after intubation, then every 5 min after block 5,10,15, and 20 min, then at skin incision, immediately after extubation, 15 min after extubation, and every 15 minutes in the post-anesthesia care unit (PACU) (30,45, and 60 minutes) till discharge of the patient.
Mean arterial blood pressure | Till discharge of the patient (Up to 12 hours)
  Mean arterial blood pressure will be recorded 5 min after intubation, then every 5 min after block 5,10,15, and 20 min, then at skin incision, immediately after extubation, 15 min after extubation, and every 15 minutes in the post-anesthesia care unit (PACU) (30,45, and 60 minutes) till discharge of the patient.
Number of doses of rescue analgesia | 12 hours after surgery
  Number of doses of rescue analgesia will be recorded.
Incidence of adverse events | 12 hours after surgery
  Incidence of adverse events will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.